CLINICAL TRIAL: NCT04306744
Title: Researching the Safety and Efficacy the Vorso PROTECT System for the Treatment of Subjects With Active Rheumatoid Arthritis Who Are naïve to Biologic or Synthetic Disease Modifying Agents
Brief Title: The RA PROTECTION Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nesos Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VC2020-7
Record Dates: First submitted 2020-03-05; First posted 2020-03-13 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, sham-controlled pilot study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Vorso PROTECT System- ON (Experimental): The subject will use the Vorso PROTECT System daily. This experimental group will have the stimulation turned on for all of the daily sessions.
  Interventions: Device: Vorso PROTECT System
- Sham Arm (Sham Comparator): The subject will use the Vorso PROTECT System daily. This experimental group will have the stimulation turned off for all of the daily sessions.
  Interventions: Device: Vorso PROTECT System - Sham (OFF)

INTERVENTIONS:
Device: Vorso PROTECT System — The Vorso PROTECT System is designed to deliver targeted, imperceptible, non-invasive stimulation to the ear to treat the signs and symptoms (e.g., tender and swollen joints, pain, synovitis) of patients with rheumatoid arthritis.
  Arms: Vorso PROTECT System- ON
Device: Vorso PROTECT System - Sham (OFF) — Identical device to experimental arm, but the device will not deliver stimulation
  Arms: Sham Arm

SUMMARY:
This is a prospective, multi-center, double-blind, randomized, controlled pilot study to assess safety and efficacy of the Vorso PROTECT System in patients who have moderately to severely active rheumatoid arthritis.

Eligible participants will be randomized in a 1:1 ratio of treatment to control (non- therapeutic) group after it has been determined they meet all of the inclusion criteria and none of the exclusion criteria. Both the treatment and control group participants will be asked to use the VORSO System once a day while maintaining a stable dose of methotrexate throughout the 12-week study. Participants will return to the site at 1, 6 and 12 weeks for follow-up testing.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 80 years of age at the time of enrollment
* Diagnosis of rheumatoid arthritis based on the 2010 EULAR/ACR criteria
* Diagnosis present for ≥3 months
* Have evidence of active disease, as defined by having at least 4 tender and 4 swollen joints in the TJC68 and SJC66, respectively
* Presence of rheumatoid factor or anti-CCP antibody at enrollment
* Must have an inadequate response to the maximum tolerated dose of 15-25 mg/week (unless lower dose is needed to due toxicity or physician discretion) of csDMARD/s for at least 12 weeks with a stable dose for at least 4 weeks prior to Baseline visit and have not been previously treated with a biologic
* Participants receiving a nonsteroidal anti-inflammatory drug (NSAID), prednisone or prednisone equivalent (10mg or less/day) or methotrexate must be on stable doses of these agents for more than 30 days prior to Baseline and remain stable for the duration of the study
* Able to operate the device appropriately and use it as per the protocol requirements
* Be willing and capable of giving informed consent
* Be willing and able to comply with research-related requirements, procedures, assessments and visits

Exclusion Criteria:

* Previously treated with any approved or investigational biologic agent (including TNF-, IL-1, IL-6, T-cell or B-cell targeted therapies) or tsDMARD
* History of any arthritis with onset prior to age 17 years or current diagnosis, inflammatory joint disease other than RA (including but not limited to gout, systemic lupus erythematosus, psoriatic arthritis, axial spondyloarthritis including ankylosing spondylitis and non-radiographic axial spondyloarthritis, reactive arthritis, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, fibromyalgia. Current diagnosis of secondary Sjogren's Syndrome is permitted.
* Participants receiving intraarticular, intramuscular, or intravenous glucocorticoids within 4 weeks prior to Baseline (unless participant is on stable dose of prednisone as per inclusion above) or if it is anticipated that the participant will need glucocorticoids at some point during the expected study duration
* Have active disease involving the auricle or ear canal (e.g. otitis media, tinnitus, infection, perforated tympanic membrane, vestibular and/or balance, excessive cerumen production), unwilling to remove a piercing (e.g. daith or tragus), or use a device (e.g. hearing aid, cochlear implant) that would preclude daily use of the earpiece
* History of any clinically significant (as deemed by PI) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, neurologic, gastrointestinal, immunologic, or other major diseases
* History of unilateral or bilateral vagotomy
* History of recurrent vasovagal syncope episodes
* Any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the research or confounds the ability to interpret data from the research in the opinion of the Investigator
* Previously implanted electrically active medical devices (e.g., cardiac pacemakers, automatic implantable cardioverter-defibrillators)
* Be pregnant or breast feeding (if female and sexually active, participant must be using a reliable form of birth control, be surgically sterile or be at least 2 years post-menopausal)
* Have symptomatic osteoarthritic knee issues within 30 days of enrollment
* Diagnosis of cancer (other than non-invasive skin cancer or carcinoma in-situ of the cervix) within the 5 years prior to research initiation
* Significant ECG findings (as determined by the Investigator), defined by:

  * Ischemic changes (defined as >1mm of down-sloping ST segment depression in at least two contiguous leads)
  * Q-waves in at least two contiguous leads
  * Clinically significant intra-ventricular conduction abnormalities (left bundle branch block or Wolf-Parkinson-White syndrome)
  * Clinically significant arrhythmias (e.g., current atrial fibrillation)
  * Bradyarrhythmias (e.g. Type I or type II block)
* Have been hospitalized for psychiatric disorder or attempted suicide within the last 12 months
* History of concurrent illness that requires hospitalization within 30 days prior to Baseline
* Have skin and vascular problems such as infected areas of skin, skin eruptions, dermatological conditions, open wounds or damaged or broken skin in the area where stimulation is planned
* Have uncontrolled hypertension or hypotension
* History or current abuse of or dependence on alcohol or drugs that would interfere with the results or adherence to research requirements based on the judgement of the Investigator
* Any clinically relevant abnormal findings in the physical exam, vital signs or laboratory tests that, in the opinion of the Investigator, may put the participant at risk
* Any language barrier that, in the opinion of the Investigator, would preclude communication and compliance with the research requirements
* Participation in another investigational trial during the 30 days prior to research initiation or during this study
* Any other household member currently participating in Vorso research or relative of site staff member
* If the investigator believes there is any reason that the participant will not be compliant with the study requirements and completion of evaluations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
ACR 20 | 12 weeks
  The percentage of participants achieving ACR 20 in the treatment vs. sham group

CONTACTS AND LOCATIONS:
Overall Officials: Alan Kivitz, MD, Principal Investigator — Altoona Center for Clinical Research
Locations (1):
- Altoona Center for Clinical Research, Duncansville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baker MC, Kavanagh S, Cohen S, Matsumoto AK, Dikranian A, Tesser J, Kivitz A, Alataris K, Genovese MC. A Randomized, Double-Blind, Sham-Controlled, Clinical Trial of Auricular Vagus Nerve Stimulation for the Treatment of Active Rheumatoid Arthritis. Arthritis Rheumatol. 2023 Dec;75(12):2107-2115. doi: 10.1002/art.42637. Epub 2023 Nov 9. PMID 37390360